CLINICAL TRIAL: NCT05278715
Title: Clinical Study of Modified Carboplatin/vincristine Chemotherapy Regimen for Visual Function Protection in Children with Optic Pathway Gliomas
Brief Title: Modified CV Regimen in Optic Pathway Glioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, Chief physician, Beijing Sanbo Brain Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 首发-2022-2-8012
Record Dates: First submitted 2022-02-17; First posted 2022-03-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Optic Glioma; Pediatric Brain Tumor, Optic Nerve Glioma
MeSH Terms: conditions — Optic Nerve Glioma | interventions — Carboplatin; Vincristine; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- optic pathway glioma (Experimental)
  Interventions: Drug: Carboplatin; Drug: Vincristine; Drug: Recombinant human endostatin

INTERVENTIONS:
Drug: Carboplatin — Dose of carboplatin is adjusted for age (over 1 year old, full dose, 220 mg/m^2; 6 months of age or less, 66 percent of the full dose; 7 to 12 months of age, 80 percent).
Drug: Vincristine — Dose of vincristine is adjusted for age (over 1 year old, full dose, 1.5 mg/m^2; 6 months of age or less, 66 percent of the full dose; 7 to 12 months of age, 80 percent). Maximum dose is 2 mg.
Drug: Recombinant human endostatin — Recombinant human endostatin (rh-ES) is administrated at a dose of 15mg daily, for 14 consecutive days every 3 weeks.

SUMMARY:
Optic pathway glioma (OPG) can result in visual deterioration. Symptomatic patients often report deficits in visual acuity (VA), visual field, visual-evoked potentials (VEPs), strabismus, proptosis, disc swelling, and other visual/neurological problems. VA itself remains one of the most important outcome measures for OPG patients, with various studies showing strong ties of VA level to overall quality of life and well-being . Maintenance of favorable VA and vision outcomes is of paramount importance in the management of OPG.

In terms of management of OPG, surgery and radiotherapy are used on a more limited basis because of location of the tumors and risk of secondary tumors, respectively. Tumor stabilization often prioritized, and chemotherapy is considered ideal for tumor stabilization in OPG, but vision is not always retained and may worsen in some cases, partially due to low radiographic efficacy and long time interval to response of the current chemotherapy regimen.

In the prior study, the investigators modified the traditional carboplatin combined with vincristine regimen by increasing the dose of carboplatin and combining with an anti-angiogenic drug. Of the 15 OPG patients, objective response rate was 80% and the time to response was only 3.3 months. 8 (53%) patients experienced an improvement in visual acuity during therapy and 6 (40%) were stable, which was higher than the historical studies.

This study was launched to further verify the clinical efficacy of the modified regimen and its effect on visual acuity improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3months and ≤21years;
* Patients with optic pathway gliomas diagnosed by histopathology or characteristic brain MRI and clinical features;
* Measurable lesions, surgical resection degree < 95% or postoperative residual tumor ≥1.5cm^2;
* KPS score ≥50 (age >12 years) or Lansky score ≥50 (age ≤12 years);
* Clinical symptoms such as decreased visual acuity, visual field defect, optic disc edema, exophthalmia, increased intracranial pressure, diencephalic syndrome, etc;
* No dysfunction of major organs.

Exclusion Criteria:

* MRI examination is not available.
* Failing to comply with the visual examination.
* H3K27 mutations, even histopathological grade 1/2.
* Receiving any other investigational agent.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the drugs used in this study.
* Patients who have received organ transplants.
* Patients infected with HIV or treponema pallidum.
* Suffering from serious cardiovascular disease;T wave inversion or elevation or ST segment changes.
* Patients who had coagulation disorder and were being treated with thrombolytic or anticoagulant drugs. Patients with significant clinical bleeding symptoms or clear bleeding tendency occurred within 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, gastrointestinal perforation, baseline fecal occult blood ++ or above, intratumoral or intracranial bleeding, or vasculitis, etc. Arteriovenous thrombosis events (such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage and cerebral infarction), deep vein thrombosis and pulmonary embolism) occurred within 6 months before enrollment.
* Pregnant or breastfeeding.
* Other conditions considered inappropriate by the researcher for inclusion.

Ages: 3 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
VA improvement rate | up to 3 years
  Percentage of visual acuity improvement

SECONDARY OUTCOMES:
time to VA improvement | up to 3 years
  Time interval from the beginning of chemotherapy to VA improvement
objective response rate | up to 3 years
  the percentage of patients who achieved confirmed complete response, partial response or minor response
median time to response | up to 3 years
  Time interval from the beginning of chemotherapy to achieving complete response, partial response or minor response

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Sanbo Brain Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No